CLINICAL TRIAL: NCT07175753
Title: The Effects of Chiropractic Applied Clinical Neuroscience Care on Sports-Related Concussion Patients: An Observational Study
Brief Title: Chiropractic Neuroscience Care in Sports Concussion
Acronym: SRC
Status: Enrolling by invitation | Type: Observational
Sponsor: Life University (Other)
Responsible Party: Sponsor
Other Study IDs: I-0033
Record Dates: First submitted 2025-07-21; First posted 2025-09-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Sports Related Concussion
Keywords: Sports related concussion; Chiropractic clinical care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SRC Group: Those who have sport-related concussion symptoms such as headache, nausea, dizziness, loss of consciousness, amnesia, balance impairment, irritability, visual disturbance, slow reaction times, etc.
  Interventions: Other: chiropractic applied clinical neuroscience care

INTERVENTIONS:
Other: chiropractic applied clinical neuroscience care — Standard chiropractic care with physiotherapy and phototherapy over two sessions

SUMMARY:
The goal of this study is to evaluate our study design and the potential effect of chiropractic-applied clinical neuroscience care on individuals with sports-related concussion (SRC) in individuals between the ages 18 and 40.The main question it aims to answer is:

- Is there any potential effect of chiropractic neuroscience care on sports related concussion patients?

Participants will be assessed on their attention, processing speed, fine motor function, standing balance, auditory function, and emotional state as part of the study using the NIH toolbox.

DETAILED DESCRIPTION:
The investigators shall recruit 20 participants for this study who are currently active athletes affiliated with the Life University Athletics Department, aged between 18 and 40 years and have sport-related concussion symptoms such as headache, nausea, dizziness, loss of consciousness, amnesia, balance impairment, irritability, visual disturbance, slowed reaction times, etc.

Subjects will do the following tasks:

1. Attention and Self-Control Test: In this test participants will look at rows of five fish on a screen and choose the direction of the middle fish while ignoring the others and press a button to show the direction of the middle fish.
2. Processing Speed Test: Participants will see two pictures side by side and decide if the pictures are the same or different and press a button as fast as they can.
3. Hand Skill Test: Subjects will be asked to do a hand skill/coordination test (called the 9-Hole Pegboard Test), where they place small pegs into holes and take them out as quickly as they can.
4. Standing Balance Test: In this test participants will stand still in various positions, sometimes with your eyes open and sometimes closed, on both hard ground and a soft foam pad, while trying to remain as still as possible. On one part of the test, they will stand with one foot in front of the other.
5. Hearing in Noise Test: Subjects will listen to words through headphones while background noise is playing. They will repeat the words they hear.
6. Emotion Surveys: They will answer questions about their feelings and relationships. These include how often they feel angry, sad, or lonely, and how happy or satisfied they feel with their life.

Assessments will be approximately 80 minutes over two sessions.

ELIGIBILITY:
Inclusion Criteria:

* Currently active athletes affiliated with the Life University Athletics Department
* Aged between 18 and 40 years
* Experiencing sport-related concussion symptoms, including but not limited to:
* Headache
* Nausea
* Dizziness
* Loss of consciousness
* Amnesia
* Balance impairment
* Irritability
* Visual disturbance
* Slowed reaction times

Exclusion Criteria:

* Not affiliated with the Life University Athletics Department
* Younger than 18 or older than 40 years
* No current symptoms of sport-related concussion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals between the ages 18 and 40 experiencing sports related concussion and symptoms such as headache, nausea, dizziness, loss of consciousness, amnesia, balance impairment, irritability, visual disturbance, slowed reaction times, etc.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-06-16 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Complete All Study Visits and Procedures | 1 year
  The number of participants who complete all scheduled study visits, tests, and treatments without early withdrawal. This measure assesses participant tolerability and compliance with the full study protocol. The unit of measure is the number of participants completing full study protocol.
Recruitment | 1 year
  Number of participant enrolled in the study within the recruitment period.
Retention | 1 year
  Number of participants who remain enrolled and complete the study protocol.
Adherence | 1 year
  Number of completed required study visits and treatments per participant.

SECONDARY OUTCOMES:
Change in Executive Function, Attention, and Inhibitory Control | 1 year
  Change from baseline in Flanker Inhibitory Control and Attention Test (FICAT) scores using the NIH Toolbox. The unit of measure is the T score on FICAT.
Change in Visual Processing Speed | 1 year
  Change from baseline in Pattern Comparison Processing Speed Test (PCPS) scores using the NIH Toolbox. The unit of measure is T score of the PCPS.
Change in Fine Motor Skills and Dexterity | 1 year
  Change from baseline in 9-Hole Pegboard Dexterity Test scores using the NIH Toolbox. Unit of measure is time in seconds to complete task (9-Hole Pegboard Test, NIH Toolbox)
Change in Postural Stability and Balance | 1 year
  Change from baseline in Balance Test scores using the NIH Toolbox Balance V3, Unit of measure is time in seconds using the NIH Toolbox Balance V3.
Change in Auditory Processing and Speech Recognition in Noise | 1 year
  Change from baseline in Words-In-Noise (WIN) Test scores using the NIH Toolbox. Unit of measure is T score from WIN Test.
Change in Negative Affect of Anger and Sadness | 1
  Change from baseline in Emotional Battery Test scores using the NIH toolbox. Unit of measure is T score of Emotional Battery Test using NIH toolbox.
Change in Emotional Support and Loneliness | 1
  Change from baseline in social relationships using Emotional Battery Test scores using the NIH toolbox. Unit of measure is T score of Emotional Battery Test.
Change in Psychological Well-being (General Life Satisfaction and Positive Affect) | 1 year
  Change from baseline in psychological well-being using the Emotional Battery Test scores using the NIH toolbox. Unit of measure is T score of Emotional Battery Test using NIH toolbox.
Acceptability from Participant Perspective | 1 year
  Participant ratings of acceptability of Sports Related Concussion intervention using a structured questionnaire. Unit of measure is the score of participants acceptability questionnaire using Likert scale (1-5) 1- Not at all, 2 - A little bit, 3 - Somewhat, 4 - Quite a bit, 5 - Very much
Acceptability from Clinician Perspective | 1 year
  Clinician ratings of acceptability of the Sports Related Concussion intervention, using a structured questionnaire. Unit of measure is the score of clinicians acceptability questionnaire using Likert scale 1- Strongly disagree, 2 - Disagree, 3 - No opinion, 4 - Agree, 5 - Strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Taha Begum, MBBS, PhD, Principal Investigator — Life University
Locations (1):
- NeuroLife Institute, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No